CLINICAL TRIAL: NCT06869980
Title: Efficacy of Limited Right Anterior Thoracotomy Versus Median Sternotomy for Mitral Valve Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB # 9413-13-4-2022
Record Dates: First submitted 2025-02-25; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-01

CONDITIONS: Minimal Invasive Cardiac Surgery; Limited Right Anterior Thoracotomy for Mitral Valve Replacement
Keywords: mitral valve replacement; Limited Right Anterior Thoracotomy; median sterntomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Limited Right Anterior Thoracotomy (Experimental): mitral valve replacement through minimal invasive approach
  Interventions: Procedure: mitral valve replacement through limited right anterior thoractomy
- median sternotomy (Active Comparator): mitral valve replacement through traditional median sterntomy approach
  Interventions: Procedure: mitral valve replacement through median sterntomy

INTERVENTIONS:
Procedure: mitral valve replacement through limited right anterior thoractomy — The incision is placed just lateral to the nipple over the fourth intercostal space (above the nipple in men and in the inframammary crease in most women) 6-10 cm in length, the pectoralis muscles are mobilized for fourth intercostal space thoracic entry-The pericardium is opened 2-cm ventral to the phrenic nerve under direct vision and carried cephalad to the aortic reflection. The anterior edge of the pericardium is tacked to incision edges using silk sutures-To initiate cardiopulmonary bypass, Cannulation of the femoral artery and femoral vein should be prior to mediastinal dissection-. The ascending aorta occluded with an external clamp. This aortic clamp passed through the thoracotomy incision if we use the aortic cross clamp and the anterograde cardioplegia delivered through a standard cardioplegia cannula secured with purse-string sutures in the ascending aorta.
  Arms: Limited Right Anterior Thoracotomy
Procedure: mitral valve replacement through median sterntomy — The incision is begun approximately 2 cm below the sternal notch and extended approximately 2 cm beyond the distal tip of the xiphoid process and is usually extended with the electrocautery down to the sternal periosteum. A midline approach can be ensured by careful attention to the insertion points of the pectoralis major muscles onto the sternum; the incision should lie directly midway between these insertion points.After sternotomy, the pericardium is opened; the heart is cannulated for cardiopulmonary bypass. Arterial inflow is established by cannulation of the distal ascending aorta near the pericardial reflection. Double venous cannulation of the venae cavae by way of the right atrium is generally employed. In most adults a size 32 Fr cannula in the superior vena cava and a size 34-38 Fr cannula in the inferior vena cava provide excellent venous drainage and easy fit. Encircling of the venae cavae and their generous mobilization aid in the subsequent exposure of the mitral valve.
  Arms: median sternotomy

SUMMARY:
this study compare between two diffrent methods for approach mitral valve in mitral valve replacement throgh opening of the middle of the sternum by saw or through opening between 4th and 5th rib on the right side of the chest without saw

DETAILED DESCRIPTION:
study the efficacy of mitral valve replacement by median sterntomy versus limited right thoractomy

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acquired isolated mitral valve disease requiring mitral valve replacement > 18 years

Exclusion Criteria:

* patients with Previous cardiac surgery, • Patients less than 18 years, • Patients with other valvular heart lesions (aortic valve or tricuspid valve) , IHD Patients , Obese patients (BMI>35), COPD patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
length of skin incision (cosmotic scar) | 1 week after surgery
  measured by centimetre by ruler
post operative pain threshold (Visual analog scale (VAS):0 to 10 assess pain from no pain-mild -moderate- sever-worst pain possible | 5 days after surgery
  measured by universal pain assessment tool
wound satisfaction scale (quality of life questionnaire) | 2 weeks after surgery
  modified Likert scale for wond satisfaction:(very dissatisfied,dissatisfied,neutral, satisfied,very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Sa Abdalla, lecturer, Principal Investigator — cardiothoracic surgery department-faculty of medecine-Zagazig univeristy-Egypt
Locations (1):
- Mohamed Samy Abdalla, Zagazig, Sharqia Province, Egypt